CLINICAL TRIAL: NCT04878887
Title: Comparaison Between Ultrasound-guided Distal and Proximal Approaches for Radial Artery Catheterization in Intensive Care Unit
Brief Title: DRA vs PRA for US-guided Radial Artery Catheterization in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Trabelsi Becem, associate professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DRA UTRAC
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Ultrasonography
Keywords: Catheter; radial artery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IP-DRA (Other): In plane distal radial artery catherterization
  Interventions: Procedure: IP-DRA vs IP- PRA
- IP-PRA (Other): In plane proximal radial artery catherterization
  Interventions: Procedure: IP-DRA vs IP- PRA

INTERVENTIONS:
Procedure: IP-DRA vs IP- PRA — Catetherization approach in plane : distal radial artery VS proximal radial artery

SUMMARY:
Patients were randomly divided into two groups: ultrasound-guided (US-guided) in-plane distal radial access (IP-DRA) and in-plane proximal radial access (IP-PRA) catheterization.

For IP-DRA , a linear transducer is placed in the radial fossa, which is known as the snuff-box. After obtaining a long-axis view of the radial artery ,the needle is inserted in the midpoint of the small footprint transducer. Then,the needle is advanced under real-time US guidance until visualizing the tip of the needle inside the artery .

For IP-PRA , a linear transducer is placed in the standard conventional forearm radial.

After obtaining a long-axis view of the radial artery ,the needle is inserted in the midpoint of the small footprint transducer. Then,the needle is advanced under real-time US guidance until visualizing the tip of the needle inside the artery .

DETAILED DESCRIPTION:
*Ultrasound-guided catheterization of the radial artery, by proximal approach:

* Patient's hand in hyperextension with slight dorsiflexion of the wrist.
* The placement of the ultrasound probe initially linear in order to obtain the "short axis" image of the artery; then a quarter turn until obtaining a longitudinal "long axis" view.
* The operator must identify the artery using the pulsed wave Doppler;
* Insertion of the needle in the middle of the transducer providing an "in plane" orientation. Thus the needle was advanced slowly and its tip was visualized throughout the procedure. *Ultrasound-guided catheterization of the radial artery, by distal approach:
* If the right hand is along the body / if the left hand is on the trunk.
* The ultrasound probe placed at the level of the anatomical snuffbox by placing the transducer in a linear fashion then rotated coronally until a longitudinal image is obtained *In the 2 groups: - The longitudinal "in plane" approach is used - After visualization of the penetration of the bevel of the needle into the lumen of the artery and the jet of arterial blood into the syringe on aspiration, a flexible metal guide was introduced into the artery through the trocar according to the Seldinger's method. - The correct positioning of the guide in the artery was then confirmed by ultrasound. Any obstacle preventing insertion of the guide system always led to a new puncture.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in intensive care unit requiring a central venous catheter (CVC)

Exclusion Criteria:

* Patients with radial AV shunt for hemodialysis
* Patients with Renaud phenomenon or lymphedema
* Congenital or acquired deformity of arms
* Cannulation site infection, hematoma and surgery

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
The overall access time | During the cannulation procedure
  Time from the ultrasound scanning to the ultrasound confirmation of the correct position of the guidewire .

SECONDARY OUTCOMES:
2. Puncture Attempts | During the procedure
  Which is the number of puncture attempts from first one until the successful one
3. The guidewire time | during the procedure
  Time from the first skin puncture to the ultrasound confirmation of the correct placement of the guidewire
4. The access time | during the procedure
  time between the first skin puncture and the jet of arterial blood
5. Rare complications | After 01 weeks of the procedure.
  Pseudo-aneurysm, AV fistula formation, radial artery dissection, which are assessed by Doppler US. In addition to radial artery eversion or perforation.

CONTACTS AND LOCATIONS:
Overall Officials: Mechaal Ben Ali, Professor, Study Chair — University Tunis El Manar
Locations (1):
- Mrezga Nabeul Tunisie, Nabeul, Tunisia

REFERENCES:
- [Background] Deepika K, Palaniappan D, Fuhrman T, Saltzmanm B. Anatomic snuffbox radial artery cannulation. Anesth Analg. 2010 Oct;111(4):1078-9. doi: 10.1213/ANE.0b013e3181ef343a. No abstract available. PMID 20870991
- [Background] Hansen MA, Juhl-Olsen P, Thorn S, Frederiksen CA, Sloth E. Ultrasonography-guided radial artery catheterization is superior compared with the traditional palpation technique: a prospective, randomized, blinded, crossover study. Acta Anaesthesiol Scand. 2014 Apr;58(4):446-52. doi: 10.1111/aas.12299. Epub 2014 Mar 3. PMID 24588456
- [Background] Kucuk A, Yuce HH, Yalcin F, Boyaci FN, Yildiz S, Yalcin S. Forty-five degree wrist angulation is optimal for ultrasound guided long axis radial artery cannulation in patients over 60 years old: a randomized study. J Clin Monit Comput. 2014 Dec;28(6):567-72. doi: 10.1007/s10877-014-9552-z. Epub 2014 Jan 11. PMID 24414382
- [Background] Sethi S, Maitra S, Saini V, Samra T, Malhotra SK. Comparison of short-axis out-of-plane versus long-axis in-plane ultrasound-guided radial arterial cannulation in adult patients: a randomized controlled trial. J Anesth. 2017 Feb;31(1):89-94. doi: 10.1007/s00540-016-2270-6. Epub 2016 Oct 19. PMID 27761661
- [Background] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Result] Pyles ST, Scher KS, Vega ET, Harrah JD, Rubis LJ. Cannulation of the dorsal radial artery: a new technique. Anesth Analg. 1982 Oct;61(10):876-8. No abstract available. PMID 7125255